CLINICAL TRIAL: NCT01453842
Title: Diet Oil Induced Stimulation of GLP-1
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Katrine Bagge Hansen, MD, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Diet oil
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glucagon-like peptide-1; Glucose-dependant insulinotropic polypeptide; Glucagon; Peptide PYY; 2-oleyl glycerol
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet; Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diet oil (Experimental)
  Interventions: Dietary Supplement: Diet oil
- Olive oil (Active Comparator)
  Interventions: Dietary Supplement: Olive oil
- Carrot (Placebo Comparator)
  Interventions: Dietary Supplement: Carrot

INTERVENTIONS:
Dietary Supplement: Diet oil — Carrot and diet oil (containing 2-OG) and 1½ g of paracetamol
  Arms: Diet oil
Dietary Supplement: Olive oil — Carrot and olive oil and 1½ g of paracetamol
  Arms: Olive oil
Dietary Supplement: Carrot — Carrot and 1½ g of paracetamol
  Arms: Carrot

SUMMARY:
Activation of G protein-coupled receptor GPR119 stimulates glucagon-like peptide-1 (GLP-1)release from the intestinal L-cells. Previously, administration of 2-oleyl-glycerol (2-OG) to humans significantly increased plasma GLP-1. In the present study we want to test the effect in patients with type 2 diabetes. The hypothesis is that we will expect to find a significant increased plasma GLP-1 following a meal containing of 2-OG when compared to meals containing of olive oil or carbohydrates alone.

DETAILED DESCRIPTION:
Activation of G protein-coupled receptor GPR119 stimulates glucagon-like peptide-1 (GLP-1)release from the intestinal L-cells. Previously, administration of 2-oleyl-glycerol (2-OG) to humans significantly increased plasma GLP-1. In the present study we want to test the effect in patients with type 2 diabetes. The hypothesis is that we will expect to find a significant increased plasma GLP-1 following a meal containing of 2-OG when compared to meals containing of olive oil or carbohydrates alone. The aim of the study is to elucidate the effect of 2-OG, 'diet oil' on GLP-1 secretion in patients with type 2 diabetes and to explain the mechanism behind the known stimulation of GLP-1 release by dietary fat.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus according to the WHO criteria
* caucasians
* age above 18 years
* BMI 20-30

Exclusion Criteria:

* kidney disease
* liver disease
* retinopathy
* anaemia
* use of insulin
* use of GLP-1 analogues
* use of DPP-4 inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Plasma GLP-1 | 3 hours
  Glp-1 response is measured during and three hours after ingestion of the different mealtest

SECONDARY OUTCOMES:
Plasma insulin | 3 hours
  Plasma insulin is measured during and 3 hours after mealtest
Plasma glucose | 3 hours
  Plasma glucose is measured during and 3 hours after meal test
Plasma GIP | 3 hours
  Plasma GIP is measured during and 3 hours after meal test
Plasma glucagon | 3 hours
  Plasma glucagon is measured during and 3 hours after meal test
Plasma PYY | 3 hours
  Plasma PYY is measured during and 3 hours after meal test
Plasma paracetamol | 3 hours
  Plasma paracetamol is measured during and 3 hours after meal test

CONTACTS AND LOCATIONS:
Overall Officials: Katrine B Hansen, MD, Study Chair — University of openhagen; Jens J Holst, Professor, Study Chair — University of Copenhagen; Harald S Hansen, Professor, Study Chair — University of Copenhagen
Locations (1):
- Department of Clinical Physiology, Glostrup Municipality, Denmark